CLINICAL TRIAL: NCT05108363
Title: Effect of Obstructive Sleep Apnea on Glucose Control and Cognitive Function - a Substudy of 'Continuous Glucose Monitoring as an Adjunct to Lifestyle Modification in Individuals With Impaired Glucose Tolerance: a Randomised Controlled Trial'
Brief Title: Effect of Obstructive Sleep Apnea on Glucose Control and Cognitive Function
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no funding
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Susanna SS Ng, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGM-OSA
Record Dates: First submitted 2021-10-24; First posted 2021-11-04 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Cognitive Change

STUDY DESIGN:
Intervention Model Description: And lifestyle modification program for 6 months of therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle modification program (Other): Patients with obstructive sleep apnea and prediabetes will have lifestyle modification program for 12 months
  Interventions: Behavioral: Lifestyle modification program

INTERVENTIONS:
Behavioral: Lifestyle modification program — Participants will attend dietary consultation sessions weekly in the first 4 months during the intensive phase , and monthly in the subsequent 8 months in the maintenance phase of LMP either face-to-face or via telephone. Participants will be given an individualized menu plan aiming at achieving a varied balanced diet with an emphasis on fiber intake and moderate-carbohydrate, low-fat, low-glycemic index products in appropriate portions. The diet will aim for a calorie reduction of 10-20%, at least 10% body weight reduction or body mass index less than 23 kg/m2.Participants will see an exercise instructor a minimum of four times starting at the 2nd month. The exercise instructor will design a suitable exercise regime. Participants will first be advised to increase daily physical activities or to do moderate intensity aerobic exercise, with the goal of 30 minutes for 3 to 5 days a week.

SUMMARY:
Obstructive sleep apnea (OSA) may contribute to altered cognitive function in patients suffering from severe OSA. And lifestyle modification program may improve the cognitive function after 6 months of therapy.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 25kg/m2
* impaired glucose tolerance which defined as plasma glucose at the range of 7.8 and 11 mmol/l 2 hours after 75g oral glucose solution intake,
* willing to participate in lifestyle modification program
* and capable of using continuous glucose monitoring (CGM) as judged by investigator

Exclusion Criteria:

1. Lactating or pregnant,
2. known diabetes, current or previous use of glucose lowering drug
3. current participation in other weight loss or lifestyle interventions, or use of weight loss drugs,
4. current use of steroids
5. uncontrolled thyrotoxicosis
6. allergy to medical grade adhesives
7. known obstructive sleep apnea on continuous positive airway pressure therapy
8. symptoms of cognitive deterioration (according to the Hong Kong Montreal Cognitive Assessment (HK-MoCA) at the score of <21)
9. predominant central sleep apnea
10. uncontrolled hypertension (blood pressure >140/90mmHg) or requiring more than two anti-hypertensive medication
11. history of stroke or brain injury,
12. unstable cardiovascular disease (e.g. recent unstable angina or myocardial infarction within the previous 6 months or severe left ventricular failure; neuromuscular disease affecting or potentially affecting respiratory muscles; moderate to severe respiratory disease (i.e. breathlessness affecting activities of daily living) or documented hypoxemia or awake SaO2 <92%)
13. psychiatric disease that limits the ability to give informed consent or complete the study
14. Use of psychoactive medication.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Change of Montreal Cognitive Assessment (MoCA) score | 12 months
  Scores on the MoCA range from zero to 30, with a score of 26 and higher generally considered normal.

SECONDARY OUTCOMES:
Change of apnea-hypopnea index | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Ng, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, China